CLINICAL TRIAL: NCT04527393
Title: Effects of Individualized Opioid Analgesia Versus Conventional Opioid Analgesia After Adenotonsillectomy in Children
Brief Title: Individualized Analgesia for Pediatric Adenotonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL-001-2020
Record Dates: First submitted 2020-08-24; First posted 2020-08-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Adenotonsillectomy; Analgesia
Keywords: adenotonsillectomy; individualized opioid analgesia; respiratory parameters; children
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individualized opioid analgesia regimen group (Experimental): The dose of oral morphine for patients in the individualized group is determined according to the results of fentanyl test.
  Interventions: Drug: Individualized oral morphine
- conventional opioid analgesia regimen group (Active Comparator): Patients in the conventional group are given routine dose of oral morphine.
  Interventions: Drug: Conventional oral morphine

INTERVENTIONS:
Drug: Individualized oral morphine — Analgesic effectiveness is assessed using the Faces Scale by the parents every four hours from postoperative Day 1 to Day 10 (eg: 8:00, 12:00, 16:00, and 20:00, each day).
  If the Faces Scale score > 6, the child receive rescue oral morphine analgesia. Patients with positive results of fentanyl test receive oral morphine 100μg/kg per dose, while patients with negative results receive oral morphine 500μg/kg per dose.
  Other Names: Individualized group
  Arms: individualized opioid analgesia regimen group
Drug: Conventional oral morphine — Analgesic effectiveness is assessed using the Faces Scale by the parents every four hours from postoperative Day 1 to Day 10 (eg: 8:00, 12:00, 16:00, and 20:00, each day).
  If the Faces Scale score > 6, the child receive rescue oral morphine analgesia. Patients receive oral morphine 200μg/kg per dose.
  Other Names: Conventional group
  Arms: conventional opioid analgesia regimen group

SUMMARY:
The objective of this randomized clinical trial is to assess the safety and effectiveness of post-adenotonsillectomy analgesia with individualized opioid analgesia regime in children.

DETAILED DESCRIPTION:
Patients will be randomly assigned to individualized opioid analgesia regimen group or conventional opioid analgesia regimen group.

Intravenous 1μg/kg fentanyl is administered as a test in patients with spontaneous breath after sevoflurane induction. A positive result is defined as a decrease of more than 50% in spontaneous respiratory rate (rate after fentanyl test versus rate before fentanyl test). Otherwise it is defined as a negative result.

All the patients are given regular paracetamol and ibuprofen after surgery. The addition of rescue oral morphine is given as needed. The dose of oral morphine is determined according to the results of fentanyl test in the individualized group, while the patients in the conventional group are given the routine dose. The Faces Scale is used to assess analgesic effectiveness by parents from postoperative day 1 to day 10. If the Faces Scale score > 6, the child receive rescue oral morphine analgesia.

At the preoperative appointment, parents are provided with a pulse oximeter including oxygen saturation sensors to take home. The oxygen saturation per night during sleep will be monitored using the pulse oximeter by parents from postoperative Day 1 to Day 10. The research team will instruct parents on how to properly apply the oximeter to the child and repeat these measurements. The primary outcome measure is desaturation events during sleep per night.

ELIGIBILITY:
Inclusion Criteria:

* Children, ASA physical status I or II, who is scheduled to undergo adenotonsillectomy will be recruited.

Exclusion Criteria:

* Children with craniofacial deformities, neuromuscular diseases, mental retardation, body mass index > 30kg/m2 , or a recent history of opioid use are excluded.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 542 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Desaturation events | from postoperative day 1 to day 10, each night
  The oxygen saturation per night during sleep will be monitored using a pulse oximeter by the parents from postoperative Day 1 to Day 10. The research team will instruct parents on how to properly apply the oximeter to the child and repeat these measurements. The primary outcome measure is desaturation events during sleep per night.

SECONDARY OUTCOMES:
Scores of Pain Scale (the Faces Scale) | every four hours from postoperative Day 1 to Day 10 (eg: 8:00, 12:00, 16:00, and 20:00, each day)
  Analgesic effectiveness was assessed using the Faces Scale by the parents every four hours from postoperative Day 1 to Day 10. Parents are trained by the research staff on how to complete pain scale.
Scores of Pain Scale (the Objective Pain Scale) | every four hours from postoperative Day 1 to Day 10 (eg: 8:00, 12:00, 16:00, and 20:00, each day)
  Analgesic effectiveness was assessed using the Objective Pain Scale by the parents every four hours from postoperative Day 1 to Day 10. Parents are trained by the research staff on how to complete pain scale.
Tonsillar bleeding events | from postoperative day 1 to day 10
  This include any signs of significant oral or nasal bleeding. It is recorded by the parents as occurring or not; if so, the number of occurrences and the time of each occurrence should be recorded.
Adverse drug reactions | from postoperative day 1 to day 10
  It is recorded by the parents as occurring or not; if so, the time of occurrence and the type of adverse reaction need to be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of Fudan university, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu HE, He L. The performance of a post-induction fentanyl-test in predicting postoperative respiratory adverse events in children after adenotonsillectomy. J Clin Sleep Med. 2024 Nov 1;20(11):1749-1754. doi: 10.5664/jcsm.11262. PMID 38935059